CLINICAL TRIAL: NCT03181009
Title: A Phase 2 Study Multi Oral Immunotherapy in Multi Food Allergic Patients to Test Immune Markers After Minimum Maintenance Dose
Brief Title: Multi OIT to Test Immune Markers After Minimum Maintenance Dose
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kari Christine Nadeau, MD PhD (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor-Investigator, Kari Christine Nadeau, MD PhD, Professor of Medicine (Pulmonary and Critical Care Medicine) and of Pediatrics (Allergy and Clinical Immunology), Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: eProtocol 39519
Record Dates: First submitted 2017-04-07; First posted 2017-06-08 (Actual); Results first posted 2019-09-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Food Allergy
Keywords: Oral Immunotherapy; Omalizumab; OIT; Xolair
MeSH Terms: conditions — Food Hypersensitivity | interventions — Omalizumab

STUDY DESIGN:
Intervention Model Description: This is a phase 2 multi site study that will be conducted at two centers in the U.S. All subjects will receive oral immunotherapy for their specific food allergies (peanut, egg, milk, wheat, soy, cashew, walnut, almond, hazelnut, sesame seed, cod, salmon and shrimp). All participants will receive three doses of Omalizumab 4 weeks apart over 8 weeks. The subject's allergens will be introduced after receiving the third omalizumab dose. Subjects will return to clinic to escalate the dose of their allergens until 300 mg (group A) vs. 1200 mg (group B) total protein daily dose is reached. There will be equivalent allergen protein portions depending on test allergen per each subject's history. Subjects will be randomized 1:1 to either group A or group B after meeting eligibility criteria. All subjects and study personnel will be blinded to group A vs B.
Who Masked: Participant, Investigator
Masking Description: Blinded labeling (Individual dosing cups will mention a choice of two doses the participant could be assigned to). Oat flour is used as the filler to create equal volumes for all doses
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (300 mg maintenance dose) (Experimental): After initial therapy with omalizumab Group A subjects will escalate their food flour allergens to 300 mg in 18 weeks.
  Interventions: Drug: Omalizumab; Drug: Food Flour Allergens
- Group B (1200 maintenance dose) (Active Comparator): After initial therapy with omalizumab Group B subjects will escalate their food flour allergens to 1200 mg in 18 weeks.
  Interventions: Drug: Omalizumab; Drug: Food Flour Allergens

INTERVENTIONS:
Drug: Omalizumab — All subjects will receive omalizumab, stored and prepared according to the investigator brochure. Subjects greater or equal to 4 yrs receive 150 mg. Subjects less than 4 yrs receive 75 mg.
  Other Names: Xolair
Drug: Food Flour Allergens — The subject's allergens will be introduced after receiving the third omalizumab dose.. Subjects will return to clinic to escalate the dose of their allergens until 300 mg (group A) vs. 1200 mg (group B) total protein daily dose is reached. There will be equivalent allergen protein portions depending on test allergen per each subject's history. Subjects will be randomized 1:1 to either group A or group B after meeting eligibility criteria. All subjects and study personnel will be blinded to group A vs B. Research staff will administer food flour to the subject orally in an age-appropriate food vehicle.
  Other Names: Food flours

SUMMARY:
Few studies have been conducted to optimize safety of multiple food allergen oral immunotherapy (OIT) in conjunction with Omalizumab as well as to identify the immunological mechanism(s) underlying any long-lasting effects of OIT. To address these issues in the field of food allergy research, we have designed this study to test whether: 1) Omalizumab improves the safety of multiple food allergen OIT in subjects with multi food allergies, 2) Omalizumab treatment with multiple food allergen OIT is associated with the ability to use a lower maintenance dose of each food allergens in the OIT regimen, particularly in younger subjects with food allergies.

DETAILED DESCRIPTION:
This is a phase 2 multisite study that will be conducted at two centers in the U.S. All subjects will receive oral immunotherapy for their specific food allergies (peanut, milk, egg, soy, wheat, cashew, walnut, almond, hazelnut, cod, salmon, sesame, shrimp). All participants will receive three doses of Omalizumab 4 weeks apart over 8 weeks. The subject's allergens will be introduced after receiving the third omalizumab dose. Subjects will return to clinic to escalate the dose of their allergens until 300 mg (group A) vs. 1200 mg (group B) total protein daily dose is reached. There will be equivalent allergen protein portions depending on test allergen per each subject's history. Subjects will be randomized 1:1 to either group A or group B after meeting eligibility criteria. All subjects and study personnel will be blinded to group A vs B.

Food protein and powder will be obtained and prepared as per Investigational New Drug 14831 and will be in compliance with all applicable regulations.

Omalizumab is approved by the European Medicines Agency (European FDA) and by the US FDA. Omalizumab will be dosed according to Genentech Dosing Omalizumab will be provided by the site.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 to 25 years with clinical history of allergy to at least two of the following: milk and/or egg and/or peanut and/or almond and/or wheat and/or cashew and/or sesame seed and/or soy and/or pecan and/or walnut and/or hazelnut and/or shrimp and/or cod and/or salmon and
* Sensitivity to food allergens documented by a positive skin prick test result greater than or equal to 6mm wheal diameter to each allergen or
* ImmunoCAP IgE level >4kU/L for each allergen and
* If female of child bearing potential, a negative urine pregnancy test before being allowed to participate in the study (week 0) and
* A plan to remain in the study area of the research center during the trial and
* Be trained on the proper use of the Epinephrine autoinjector and agree to follow epi training to be allowed to enroll in the study and
* If female of child-bearing potential, willing to be compliant with a medically-approved method of contraception (please see Pregnancy section in this IND document) and
* Agree to eliminate other known food allergens from subject's diet so as not to confound the safety and efficacy data from the study and
* Avoid open or blinded food challenges to food allergens

Exclusion Criteria:

* Previous anaphylactic reaction to Omalizumab
* A history of severe anaphylaxis to food allergens that will be desensitized in this study requiring intubation or admission to an ICU, frequent allergic or non-allergic urticaria, or history consistent with poorly controlled persistent asthma
* Unstable angina, significant arrhythmia, uncontrolled hypertension, chronic sinusitis, or other chronic or immunological diseases that, in the judgment of the investigator, might interfere with the evaluation or administration of the test drug or pose additional risk to the subject (e.g., gastrointestinal or gastroesophageal disease, chronic infections, scleroderma, hepatic and gallbladder disease, chronic non-allergic pulmonary disease)
* An average forced expiratory volume at one second (FEV1) or peak expiratory flow rate (PEF) less than 80% predicted (moderate persistent asthma) with or without controller medication (if able to perform the maneuver) at screening, or a food challenge visit
* Current users of oral, intramuscular, or intravenous corticosteroids, tricyclic antidepressants, or are taking a beta-blocker (oral or topical)
* Routinely using medication that could induce adverse gastrointestinal reactions during the study
* Refusing to sign or follow the Epinephrine autoinjector Training Form
* Pregnant or breast feeding women
* Unwilling to avoid other allergens outside this study
* Concurrent/prior use of immunomodulatory therapy (within 6 months)
* A diagnosis of eosinophilic esophagitis, eosinophilic colitis, or eosinophilic gastritis.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kari C Nadeau, MD PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - UCLA, Los Angeles, California
  - Sean N. Parker Center for Allergy and Asthma Research at Stanford, Mountain View, California

IPD SHARING:
Plan to Share IPD: Undecided
pending

REFERENCES:
- [Derived] Sindher SB, Kumar D, Cao S, Purington N, Long A, Sampath V, Zedeck SS, Woch MA, Garcia-Lloret M, Chinthrajah RS. Phase 2, randomized multi oral immunotherapy with omalizumab 'real life' study. Allergy. 2022 Jun;77(6):1873-1884. doi: 10.1111/all.15217. Epub 2022 Jan 24. PMID 35014049
- See also: Sean N. Parker Center for Allergy and Asthma Research — http://med.stanford.edu/allergyandasthma
- See also: Research Registry for the Sean N. Parker Center for Allergy and Asthma Research — http://is.gd/snpregistry

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A (300 mg Maintenance Dose) | Group B (1200 Maintenance Dose)
Started | 30 | 30
Completed | 30 | 28
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: Sixty-five participants were initially screened for eligibility with 60 ultimately randomized 1:1 to the 300 mg and 1200 mg arms at two sites. Two participants withdrew early and 11 did not reach maintenance, but continued in the study throughout duration.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (300 mg Maintenance Dose) | Group B (1200 Maintenance Dose) | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Median (Full Range); unit: years] | 10 [4 to 20] | 10 [4 to 17] | 10 [4 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 21 | 20 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 28 | 28 | 56
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60
Total IgE [Median (Full Range); unit: IU/mL] | 648 [64 to 6538] | 701 [61.00 to 4367] | 665.00 [61 to 6538.00]

OUTCOME MEASURES:

1. Primary Outcome: Change in Allergen-specific Serum IgG4 and IgE
Description: Change in allergen-specific serum IgG4 and IgE from baseline to Week 18 (End of Study)
Time Frame: 18 weeks
Measure: Median (Full Range); unit: Total serum IgE (kU/L)
Arm/Group | Group A (300 mg Maintenance Dose) | Group B (1200 Maintenance Dose)
Number analyzed (Participants) | 30 | 30
Total serum IgE (kU/L) | 578.5 [64.6 to 6538] | 738.5 [61.0 to 4367]

ADVERSE EVENTS:
Time Frame: 18 weeks
Arm/Group | Group A (300 mg Maintenance Dose) | Group B (1200 Maintenance Dose)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 19/30 | 16/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (300 mg Maintenance Dose) (N=30) | Group B (1200 Maintenance Dose) (N=30)
Abdominal pain (Gastrointestinal disorders) | 14 | 12 — nausea or vomiting
chills, facial edema, fatigue (General disorders) | 3 | 12
cough, sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
pruritus, rash (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Statistical Analysis Plan (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/09/NCT03181009/SAP_001.pdf
  • Informed Consent Form (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT03181009/ICF_002.pdf
  • Study Protocol (2017-05-23): https://cdn.clinicaltrials.gov/large-docs/09/NCT03181009/Prot_003.pdf